CLINICAL TRIAL: NCT02764086
Title: INTENSE: A Phase I/II Study of INhomogeneous Targeted Dose Escalation in Non-Small CEll Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Accrual lower than anticipated and not expected to improve
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 15-47
Record Dates: First submitted 2016-04-21; First posted 2016-05-06 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: This is a prospective non-randomised Phase I/II study with patients recruited to escalated dose cohorts. Escalated dose to the iGTV (internal gross tumour volume), with 60 Gy to the conventional PTV (planning target volume), will be delivered to successive cohorts of participants (6-12 participants/cohort) until the maximum tolerated oesophageal dose is determined. The minimum dose delivered to the iGTV will be 65 Gy, with 60 Gy to the PTV, delivered via intensity modulated radiation therapy (IMRT) or volume modulated arc therapy (VMAT), planned on an Average Intensity Projection (AVIP) dataset.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trial Cohort Description (Other): Escalated dose of min 65Gy to the iGTV, with 60Gy to PTV delivered to successive cohorts of patients(pts) until the MTD oesophageal dose is determined. Toxicity will be analysed 2 months post 6pts treated in a cohort.
  If: ≤2pts have ≥G3 toxicity, next cohort will be enrolled & receive escalated dose (an additional +5Gy at each escalation upto max 75Gy)/3 of 6pts have ≥G3 toxicity, a further 6pts will be recruited into that dose level/≥4pts have ≥G3 toxicity, the MTD is fixed at dose level of previous cohort
  Cohort is extended to 12pts:
  If: ≤4pts have ≥G3 toxicity, next cohort will be enrolled & receive escalated dose/5 of 12pts have ≥G3 toxicity, the MTD is fixed at that dose level & recruitment continues up to 24pts/≥6pts have ≥G3 toxicity, the MTD is fixed at the dose level of previous cohort.
  Once the max dose cohort is established, recruiting will continue at that dose until 24pts. Concurrent & neo-adjuvant/no chemotherapy arms will be escalated independently of each other
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Escalated dose of minimum 65Gy to the iGTV, with 60 Gy to PTV.

SUMMARY:
This is a prospective non-randomised Phase I/II study with patients recruited to escalated dose cohorts. Escalated dose to the iGTV (internal gross tumour volume), with 60 Gy to the conventional PTV (planning target volume), will be delivered to successive cohorts of participants (6-12 participants/cohort) until the maximum tolerated oesophageal dose is determined. The minimum dose will be 60 Gy delivered via intensity modulated radiation therapy (IMRT) or volume modulated arc therapy (VMAT), planned on an Average Intensity Projection (AVIP) dataset.

Standard of care chemotherapy.

There will be two treatment arms; one with patients who are planned to receive neo-adjuvant or no chemotherapy, and the other with patients who are planned to receive concurrent chemotherapy.

DETAILED DESCRIPTION:
This is a prospective non-randomised Phase I/II cohort study; please see above for Radiation Therapy and Chemotherapy treatment details

Each cohort will require a minimum of 6 and a maximum of 12 patients. Once 6 patients have been treated in a cohort a two-month break is taken before toxicity is analysed.

* If 2 or fewer patients experience a grade ≥3 toxicity, the next cohort will be enrolled and will receive an escalated dose (an additional +5 Gy at each escalation up to a maximum of 75 Gy)
* If 3 of the 6 patients experience a grade ≥3 toxicity, a further 6 patients will be recruited into that dose level
* If 4 or more patients experience a grade ≥3 toxicity then the MTD is fixed at the dose level of the previous cohort

If the cohort is extended to 12 patients, the following rules apply:

* If 4 or fewer patients experience a grade ≥3 toxicity, the next cohort will be enrolled and will receive an escalated dose.
* If 5 of the 12 patients experience a grade ≥3 toxicity, then the MTD is fixed at that dose level and recruitment continues up to a total of 24 patients at that dose level.
* If 6 or more patients experience a grade ≥3 toxicity, then the MTD is fixed at the dose level of the previous cohort.

Once the maximum dose cohort is established, patients will continue to be recruited at that dose level up to a total of 24 patients.

There will be two treatment arms; one with patients who are planned to receive neo-adjuvant or no chemotherapy, and th eother with patients who are planned to receive concurrent chemotherapy.

The concurrent and neo-adjuvant /no chemotherapy arms will then be escalated independently of each other.

For each arm the following number of patients will be required:

* Minimum number (if maximum dose level reached) = 36 (6 at 65 Gy, 6 at 70 Gy and 24 at 75 Gy)
* Maximum number (if maximum dose level reached) = 48 (12 at 65 Gy, 12 at 70 Gy and 24 at 75 Gy) A maximum of 48 patients are required to complete each arm (neo-adjuvant or none /concurrent chemotherapy) of the trial.

Acute toxicity will be assessed weekly during treatment and at 2, 4 and 8 weeks post-treatment Late toxicities will be assessed at 3, 6, 9, 12, 18 and 24 months post-treatment and annually thereafter until disease relapse / patient withdrawal / patient death.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age
2. ECOG (European Cooperative Oncology Group) performance status 0-2 (0-1 for concurrent chemotherapy)
3. Weight loss <10% within 3 months of diagnosis
4. Histological diagnosis (biopsy or cytology) of NSCLC (Squamous Cell Carcinoma (SCC), Adenocarcinoma, Large Cell).

   Eligible NSCLC stages: IIA (provided N1); IIB (including T3N0 if unresectable or unsuitable for stereotactic ablative body radiation therapy (SABR)); IIIA and IIIB
5. Inoperable (as per Multi-Disciplinary Team (MDT)) or patient refuses surgery
6. Respiratory function:

   Forced Expiratory Volume (FEV1) ≥ 1L or ≥ 40% of predicted Diffusing Capacity of Lung for Carbon Monoxide (DLCO) ≥ 40%
7. Radiological confirmation of disease via a Positron Emission Tomography (PET) scan prior to registration.
8. Life expectancy, from causes other than lung cancer, of greater than 12 months (as per physician's opinion)
9. Females of child bearing potential (see Appendix H) must not be pregnant and must be prepared to use adequate contraception methods during treatment. Males whose female partners are of child-bearing potential must be prepared to use adequate contraception methods during treatment. Examples of effective contraception methods are a condom or a diaphragm with spermicidal jelly, or oral, injectable or implanted birth control.
10. Provision of written consent in line with ICH-GCP guidelines

Exclusion Criteria:

1. Previous thoracic radiation therapy
2. Known co-existing or prior malignancy which is likely to interfere with treatment or assessment of outcomes
3. Known distant metastases or metastatic pleural effusion
4. Pancoast tumours (tumour of the pulmonary apex)
5. Supraclavicular nodal involvement
6. Spinal cord involvement
7. Patients with syndromes or conditions associated with increased radiosensitivity or development of lung fibrosis
8. Suitable for SABR
9. Idiopathic pulmonary fibrosis/usual interstitial pneumonia
10. Uncontrolled intercurrent illness that is likely to interfere with treatment or assessment of outcomes
11. Psychiatric illness/social situations that would limit compliance with study requirements
12. Pregnant or lactating at the time of proposed randomisation
13. Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study, or if it is felt by the research / medical team that the patient may not be able to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

PRIMARY OUTCOMES:
To assess the safe delivery of an achievable level of dose escalation in a dose escalated and intensified RT regime delivered via VMAT/IMRT and focused on the GTV by the proportion of grade ≥3 toxicities determined to be related to RT | 4 years 3 months

SECONDARY OUTCOMES:
To compare grade ≥3 toxicity 3, 6, 9, 12, 18 and 24 months, post-treatment, graded by NCI-CTCAE Version 4 (V4) | 2 years post treatment
To estimate the rate of overall survival; death from any cause is considered an event | 8 years
To estimate the rate of disease-free survival. All disease recurrences will be recorded. In disease-free survival, any tumour recurrence, development of distant metastases or death is considered an event. | 8 years
To estimate the time to local failure (failure defined by RECIST V1.1 ) | 8 years
To evaluate tumour response at 6, 12 and 24 months (response measured by RECIST V1.1) | 2 years
The estimate the time to distant metastases as assessed by imaging or biopsy | 8 years
To assess Quality of life according to the EORTC QLQ-C30 and EORTC QLQ-LC13 | 8 years
To assess the MTD to the oesophagus. The MTD is defined as the highest dose that does not cause unacceptable toxicities. Toxicities of interest are any CTCAE V4 grade ≥3 oesophageal toxicity determined to be related to radiation therapy. | 5 years
The change in pulmonary function post-treatment will be analysed by calculating the differences in measurements from baseline to the 1-year follow-up | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prof John Armstrong, Principal Investigator — St Luke's Radiation Oncology Network
Locations (1):
- St Lukes Radiation Oncology Network (SLRON) at St Luke's Hospital and St James Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided